CLINICAL TRIAL: NCT04158440
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase III Clinical Study on Toripalimab Combined With Platinum-Based Doublet Drug Chemotherapy for Resectable, Stage II-III, Non-Small Cell Lung Cancer
Brief Title: Phase III Study of Toripalimab Versus Placebo Plus Chemotherapy in Resectable NSCLC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-029-III-NSCLC
Record Dates: First submitted 2019-11-01; First posted 2019-11-08 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Stage II-III Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; Docetaxel

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4cycles(Toripalimab IV 240mg + platinum-based doublet chemotherapy)+13 cycles(Toripalimab IV 240mg) (Experimental): Participants receive totally 4 cycles of Toripalimab combined with platinum doublet chemotherapy during perioperative period ;After surgery, participants receive consolidation therapy of Toripalimab
  Interventions: Drug: 4cycles(Toripalimab IV 240mg + platinum-based doublet chemotherapy)+13 cycles(Toripalimab IV 240mg); Biological: Toripalimab
- 4cycles(Placebo + platinum-based doublet chemotherapy)+13 cycles(Placebo ) (Active Comparator): Participants receive totally 4 cycles of Placebo combined with platinum doublet chemotherapy during perioperative period ;After surgery, participants receive consolidation therapy of Placebo
  Interventions: Drug: 4cycles(Placebo + platinum-based doublet chemotherapy)+13 cycles(Placebo )

INTERVENTIONS:
Drug: 4cycles(Toripalimab IV 240mg + platinum-based doublet chemotherapy)+13 cycles(Toripalimab IV 240mg); Biological: Toripalimab — Biological: Toripalimab 240 mg by IV infusion every 3 weeks (Q3W), given on cycle day 1;Drug: Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1;Drug: Corboplatin AUC 5 by IV infusion Q3W, given on cycle day 1;Drug: Pemetrexed 500 mg/m^2 by IV infusion Q3W, given on cycle day 1. Given only to participants with nonsquamous NSCLC.Drug:Paclitaxel 175 mg/m^2 by IV infusion Q3W;Drug:Docetaxel 60-75 mg/m^2 by IV infusion Q3W
  Other Names: Cisplatin;; Carboplatin;; Pemetrexed;; Paclitaxel;; Docetaxel
  Arms: 4cycles(Toripalimab IV 240mg + platinum-based doublet chemotherapy)+13 cycles(Toripalimab IV 240mg)
Drug: 4cycles(Placebo + platinum-based doublet chemotherapy)+13 cycles(Placebo ) — Biological: Placebo by IV infusion every 3 weeks (Q3W), given on cycle day 1;Drug: Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1;Drug: Corboplatin AUC 5 by IV infusion Q3W, given on cycle day 1;Drug: Pemetrexed 500 mg/m^2 by IV infusion Q3W, given on cycle day 1. Given only to participants with nonsquamous NSCLC.Drug:Paclitaxel 175 mg/m^2 by IV infusion Q3W;Drug:Docetaxel 60-75 mg/m^2 by IV infusion Q3W
  Other Names: Cisplatin;; Carboplatin;; Pemetrexed;; Paclitaxel;; Docetaxel
  Arms: 4cycles(Placebo + platinum-based doublet chemotherapy)+13 cycles(Placebo )

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center, phase III clinical study to evaluate the efficacy and safety of Toripalimab injection (JS001) combined with platinum-based doublet drug chemotherapy versus placebo combined with platinum-based doublet drug chemotherapy for subjects with resectable, stage II-III NSCLC.

DETAILED DESCRIPTION:
Subjects who meet all the inclusion criteria but do not meet any exclusion criteria are randomized into two groups at a ratio of 1:1: according to the stratification factors as below:

* Disease stage: II vs IIIA vs IIIB
* PD-L1 status: PD-L1 expression ≥1% vs. PD-L1 <1% or not evaluable
* Planned surgical operation: pneumonectomy vs. lobectomy
* Pathological type: non-squamous cell carcinoma vs. squamous cell carcinoma Neoadjuvant therapy should be started within 3 days after randomization. Toripalimab IV 240 mg Q3W /plaecbo will be given combined with platinum-based doublet drug chemotherapy for three cycles in the preoperative neoadjuvant therapy period for trial group; Every 3 weeks of treatment is regarded as one cycle, in which combined therapy is given in the first day of every cycle.

All the subjects will receive preoperative radiological and surgical evaluation 3-5 weeks after neoadjuvant therapy.

After 3 cycles of preoperative neoadjuvant therapy, all the subjects who still have surgical indications will receive radical excision based on the surgical operation criteria of the World Association for Lung Cancer Research within 4-6 weeks after 3 cycles of preoperative neoadjuvant therapy. The pTNM will be staged in accordance with AJCC Cancer Staging Manual (version 8). All the specimens taken during the operation will be evaluated by local pathologists for the surgical margin. The tumor tissue samples collected from subjects during the study will be submitted to the authorized central laboratory for blinded evaluation of pathological response and translational research.

All the subjects who have completed the radical operation will receive one cycle of postoperative adjuvant therapy, i.e., Toripalimab IV 240 mg/placebo + platinum-based doublet drug chemotherapy in 30 days after the operation. If there is no adjuvant radiotherapy plan, it will proceed to consolidation treatment period three weeks after adjuvant therapy; if adjuvant radiotherapy is planned then the consolidation treatment period will start 30 days after adjuvant radiotherapy. In the consolidation treatment period, Toripalimab IV 240 mg/placebo is given in each cycle of every 3 weeks for a total of 13 cycles . Adverse events (AEs) will be monitored throughout the study, and the severity will be graded to the guidelines listed in National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0 or above. The safety will be followed up in the subjects who have received study treatment and discontinued the drug prematurely. All the subjects will be followed up for overall survival, until death, withdrawal of informed consent or end of study.

ELIGIBILITY:
Inclusion criteria：

1. Having sufficient understanding of this study and being willing to sign the informed consent form (ICF);
2. Aged 18-70 years, male or female;
3. Treatment-naive, histologically confirmed resectable, stage II, IIIA, IIIB (N2) (AJCC staging system, version 8) NSCLC; cTNM stage can be confirmed through PET-CT or pathological biopsy; resectable stage II non-small cell lung cancer is defined as eligible for radical resection evaluated by a qualified thoracic surgeon; resectable stage III is defined as the resectable and potential resectable according to the Chinese expert consensus on the multidisciplinary diagnosis and treatment for stage III non-small cell lung cancer (2019)in which resectable includes IIIA(N0-1), partial N2 with single-station mediastinal lymph node metastasis and the short diameter of lymph node<2 cm， partial T4 (satellite nodules in the adjacent lobe) N1 and potential resectable includes partial stage IIIA and IIIB with the short diameter of single-station N2 mediastinal lymph node<3 cm, other potentially resectable T3 or T4 central tumor ; Any suspected lesions which could change the TNM stage, such as contralateral mediastinal lymph node, supraclavicular lymph mode, solid/sub-solid pulmonary node and non-isolated ground glass opacity (GGO), pathological confirmation is strongly recommended.
4. Measurable lesions based on the response evaluation criteria in solid tumors version 1.1;
5. Tumor tissue specimens available for pathological diagnosis, detection of PD-L1 expression and biomarkers prior to randomization (the tumor tissue specimens must be freshly obtained or archived samples within 3 months prior to enrollment; tumor tissue specimens must be the samples of histological category, including but not limited to the tissue punctured by core needle and hollow needle, tissue acquired by bronchoscopic clamp, surgically resected samples; the samples acquired by fine needle puncture and bronchial brushing are not acceptable);
6. ECOG score 0-1;
7. Good organ function:
8. Being willing and able to comply with the visits, treatment plan, laboratory examinations and other study procedures scheduled in the study;
9. pulmonary function test being able to withstand the planned pneumonectomy evaluated by surgeons; Women of childbearing potential must undergo serum pregnancy test within 3 hours prior to the first dose and the result must be negative. Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to use highly effective contraceptive methods during the study period and within 180 days after the last dose of study drug.
10. Women of childbearing potential must undergo serum pregnancy test within 3 days prior to the first dose and the result must be negative. Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to use highly effective contraceptive methods during the study period and within 180 days after the last dose of study drug

Exclusion criteria：

1. Presence of locally advanced, unresectable or metastatic disease; unresectable includes the unresectable defined in the Chinese expert consensus on the multidisciplinary diagnosis and treatment for stage III non-small cell lung cancer (2019), including partial stage IIIA and IIIB and all the stage IIIC; N2: single station mediastinal lymph node metastasis with short diameter ≥3cm; N2: multiple station mediastinal lymph node metastasis with lymph node fusion and the short diameter of lymph node ≥2cm on CT; ALL the N3; T4: invading esophagus, heart, aorta;
2. NSCLC involving superior sulcus, large cell neuroendocrine carcinoma (LCNEC), sarcomatoid tumor;
3. Participants with known EGFR sensitive mutations or ALK translocation, EGFR and ALK mutation status needs to be identified for the subjects with non-squamous cell carcinoma;
4. Previous treatment with systemic antitumor therapy for early NSCLC, including investigational product;
5. History of (non-infectious) pneumonitis/interstitial lung disease requiring steroid treatment, or ongoing pneumonitis/interstitial lung disease requiring steroid treatment;
6. Active tuberculosis;
7. Active infection requiring systemic treatment;
8. Subjects with any known or suspected autoimmune disorder or immunodeficiency, with the following exceptions: hypothyroidism, hormone therapy is not needed, or well controlled at physiological dose; controlled type I diabetes;
9. Uncontrolled active hepatitis B (defined as positive hepatitis B surface antigen [HBsAg] in screening period with HBV-DNA detected higher than the upper limit of normal at the clinical laboratory of the study center); (the subjects with HBV-DNA assay <500 IU/mL within 28 days prior to randomization who have received local standard antiviral therapy for at least 14 days and are willing to receive antiviral therapy continuously during the study can be enrolled); active hepatitis C (defined as positive hepatitis C surface antibody [HCsAb] in screening period and positive HCV-RNA);
10. Known human immunodeficiency virus (HIV) infection (known positive HIV antibody);
11. Vaccination of live vaccine within 30 days prior to the first dose. Including but not limited to the following: parotitis, rubella, measles, varicella/ herpes zoster (varicella), yellow fever, Rabies, Bacille Calmette-Guérin (BCG) and typhoid vaccine (inactivated virus vaccine allowed);
12. ≥ Grade 2 peripheral neuropathy;
13. Previous use of PD-1/PD-L1 agent or the drug acting on another targeted T cell receptor (e.g., CTLA-4, OX-40);
14. Severe allergic reaction to other monoclonal antibodies;
15. History of serious allergy to Pemetrexed, paclitaxel or docetaxel, cisplatin, carboplatin or its preventive medications;
16. Known serious or uncontrolled pre-existing diseases; including but not limited to cardiovascular events with hemodynamic instability, symptomatic cerebrovascular events, and hepatic cirrhosis above Child-Pugh A within 6 months;
17. History or current evidence of any disease, therapy or abnormal laboratory examination that may confuse the study results, interfere with subject's participation in the full course of the study or not meet the best interest of subject's participation in the study, as judged by investigators;
18. Other malignant tumors within 5 years prior to the first dose, except non-small cell lung cancer. The malignant tumors with negligible risk of metastasis or death (e.g., expected disease-free survival > 5 years) and expected to achieve radical outcomes after treatment (e.g., sufficiently treated carcinoma in situ of cervix, basal or squamous cell skin cancer, ductal carcinoma in situ treated for radical surgery) can be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MPR rate in stage III population evaluated by BIPR | up to 7 weeks after neoadjuvant
  Major Pathological Response (MPR) Rate.MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy.
EFS in stage III population evaluated by investigators | up to 3 years
  Event Free Survival (EFS):EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause.
MPR rate in stage II-III population evaluated by BIPR | up to 7 weeks after neoadjuvant
  Major Pathological Response (MPR) Rate.MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy.
EFS in stage II-III population evaluated by investigators | EFS: up to 3 years
  Event Free Survival (EFS):EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause.

SECONDARY OUTCOMES:
pCR rate in stage III population evaluated by BIPR and investigators | pCR:up to 7 weeks after neoadjuvant;
  Pathological Complete Response (pCR) Rate :pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
EFS in stage III population evaluated by IRC | EFS by IRC:up to 3 years
  EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined either by biopsy assessed by blinded central pathologist or by imaging using RECIST 1.1 assessed by investigator.
Disease-free survival (DFS) in stage III evaluated by IRC and investigators | DFS:up to 3 years
  DFS is defined as the time from postoperation until radiographic disease progression, local or distant recurrence, or death due to any cause.
pCR rate in stage II-III population evaluated by BIPR and investigators | pCR:up to 7 weeks after neoadjuvant
  Pathological Complete Response (pCR) Rate :pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.
EFS in stage II-III population evaluated by IRC | EFS by IRC:up to 3 years
  EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined either by biopsy assessed by blinded central pathologist or by imaging using RECIST 1.1 assessed by investigator.
Disease-free survival (DFS) in stage II-III population evaluated by IRC and investigators | DFS:up to 3 years
  DFS is defined as the time from postoperation until radiographic disease progression, , local or distant recurrence, or death due to any cause.
Overall survival (OS) rate in stage III and II-III population | OS up to 5 years
  OS is defined as the time from randomization until death from any cause.
2-3 years overall survival (OS) rate in stage III and II-III population | OS up to 5 years
  OS rate is defined as survival probability n stage III and II-III population at a given time point（2y，3y）

OTHER OUTCOMES:
Safety evaluation of subjects | Safety: 90 days after the last administration
  Safety: adverse event (AE), abnormal laboratory examination, serious adverse event (SAE) related with the study drug judged using NCI-CTCAE V5.0; surgical feasibility: percentage of procedure delay or cancellation, change of surgical approach, operation time；
Exploratory analysis of potential biomarkers related with the outcome | Exploratory :withdrawal from study treatment，up to 71 weeks
  Exploratory analysis of potential biomarkers related to the outcome (including PD-L1 expression in tissue specimen, tumor mutation burden (TMB), whole exome sequencing (WES) and change of ctDNA in peripheral blood sample)
Pharmacokinetics: plasma concentration of Toripalimab in each cycle; | Exploratory : withdrawal from study treatment，up to 71 weeks
  Pre-dose serum samples will be collected from subjects at cycles 1, 2, and 3 of the neoadjuvant therapy period, cycle 1 of the adjuvant therapy period, and cycles 1, 5, 9, and 13 of the consolidation therapy period for the determination of Toripalimab concentrations.
mmunogenicity: the incidence and titer of anti-drug antibody (ADA) and whether it is neutralizing antibody (if necessary); | Exploratory : withdrawal from study treatment，up to 71 weeks
  Pre-dose serum samples will be collected from subjects at cycles 1, 2, and 3 of the neoadjuvant therapy period, cycle 1 of the adjuvant therapy period, and cycles 1, 5, 9, and 13 of the consolidation therapy period to detect the presence of anti-drug antibodies (ADAs). ADA-positive samples will be tested and analyzed for neutralizing antibodies (if necessary).

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Yes

REFERENCES:
- [Derived] Lu S, Zhang W, Wu L, Wang W, Zhang P; Neotorch Investigators; Fang W, Xing W, Chen Q, Yang L, Mei J, Tan L, Sun X, Xu S, Hu X, Yu G, Yu D, Yang N, Chen Y, Shan J, Xing L, Tian H, Zhang X, Zhou M, Fang H, Wu G, Liu Y, Ye M, Cao L, Jiang J, Li X, Zhu L, Li S, Kang M, Zhong A, Chen K, Wu N, Sun Q, Ma H, Cai K, Wang C, Lin G, Zhu K, Zhang Y, Zhang X, Hu H, Zhang W, Chen J, Yang Z, Hang X, Hu J, Huang Y, Zhang Z, Zhang L, Zhang L, Liu L, Lin D, Zhang J, Chen G, Li Y, Zhu L, Wang W, Yu W, Cao D, Keegan P, Yao S. Perioperative Toripalimab Plus Chemotherapy for Patients With Resectable Non-Small Cell Lung Cancer: The Neotorch Randomized Clinical Trial. JAMA. 2024 Jan 16;331(3):201-211. doi: 10.1001/jama.2023.24735. PMID 38227033